CLINICAL TRIAL: NCT01348711
Title: Placental Insufficiency Screening During First Trimester by a Combination of Uterine Artery Dopppler, Maternal PlGF and sFLT-1 in Hight Risk Population
Brief Title: Early Placental Insufficiency Screening
Acronym: BIODOP-T1
Status: Terminated | Type: Observational
Why Stopped: Shortness inclusions of patients
Sponsor: University Hospital, Tours (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHRI/06/FP-BIODOP-T1
Record Dates: First submitted 2010-02-02; First posted 2011-05-05 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Pre-eclampsia
Keywords: Pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — SERUM
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To assess the role of uterine artery and maternal serum PlGf and sflt-1 and their combination in screening for pre-eclampsia and small -for-gestational age (SGA) fetuses at 12-14 weeks of gestation

DETAILED DESCRIPTION:
Pre-eclampsia (PE) and intrauterine growth restriction (IUGR) are known as major factors in perinatal morbidity and mortality. Routine antenatal care is focused on the detection of women at increased risk to apply this population a program of careful monitoring and appropriate intervention.

Uterine artery Doppler during anomaly scan at 12 to 14 weeks in selected women at increased risk, has proved to be accurate to detect those who will develop PE or IUGR during the second half of pregnancy.

A variety of angiogenic proteins have been studied as potential markers for pre-eclampsia. Among these protein Plgf and sflt-1 have respectively demonstrated higher and lower levels in pregnant women who will subsequently develop pre-eclampsia.

Our study is aimed to evaluate the performance of serum Plgf and sflt-1 measurement in association with uterine artery Doppler as a screening for placental insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hypertension under medication
* Insulin or not insulin dependant preexisting diabetes
* Previous history of pre-eclampsia
* Previous history of unexplained stillbirth
* Previous history of placental abruption
* Previous history of SGA (< 10th centile)
* History of pre-eclampsia or chronic hypertension before 45 years in the mother or a sister
* History of vascular pathology before 50 years in the father
* Obesity (BMI>26)
* Nulliparous after 38 years
* Assisted conception with donor
* Primipaternity after 38 years old or before 20 years old

Exclusion Criteria:

* Multiple pregnancy
* Pregnancy requiring termination
* Unability to understand the study
* Thrombophilia
* treatment with heparin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant between 12 and 14 weeks
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2007-05; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Occurrence for Pre-eclampsia or SGA | During pregnancy and until 72h after delivery
  Pre-eclampsia is defined as hypertension (systolic blood pressure 140mmHg or greater or a diastolic blood pressure 90mmHg or greater on at least 2 occasions 4 hour or 1 week apart) accompanied by proteinuria (more or equal to 0.5g/day or 1 dipstick of ++ or more). SGA is defined as birth weight below the 10th centile for gestational age at birth according to the national birthweight distribution of the french population (INSERM)

SECONDARY OUTCOMES:
Early onset pre-eclampsia | During pregnancy and until 72h after delivery
  Early onset pre-eclampsia is defined as pre)eclampsia occurring before 32 completed gestational weeks.
Severe pre-eclampsia | During pregnancy and until 72h after delivery
  Severe pre-eclampsia is defined as systolic blood pressure of 160mmHg or greater or a diastolic blood pressure of 110mmHg or greater and/or proteinuria greater than 5g in 24 hour collection or occurrence of abruption, eclampsia (seizures during pre-eclampsia), HELLP syndrome (hemolysis, elevated enzyme liver, low platelets), renal insufficiency, fetal demise or birth weight below the 5th centile for gestational age.

CONTACTS AND LOCATIONS:
Overall Officials: Franck PERROTIN, MD-PHD, Study Director — Univsersity Hospital of TOURS
Locations (4):
- France (4):
  - Hospital of Blois -Service de Gynécologie-Obstétrique, Blois
  - CHRU Hôpital Hôtel-Dieu Département Gynécologie Obstétrique, Nantes
  - Hôpital La Milétrie, CHRU Poitiers, Poitiers
  - Olympe de Gouges Women Health Centre, Bretonneau University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No